CLINICAL TRIAL: NCT00347607
Title: Cost-effectiveness of Three Alternative Azithromycin Treatment Strategies for Trachoma Control in Tanzania
Brief Title: Study of Three Alternatives for Mass Treatment in Trachoma Villages of Tanzania
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: International Trachoma Initiative (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITI01-033
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2002-03

CONDITIONS: Trachoma
Keywords: trachoma; chlamydia trachomatis; surveillance; azithromycin
MeSH Terms: conditions — Trachoma

INTERVENTIONS:
Behavioral: community surveillance and re-treatment

SUMMARY:
After single, yearly, mass treatment of communities with azithromycin for active trachoma, what is the added effectiveness for reduction of trachoma and ocular C. trachomatis infection at one, two, and three years, relative to the added costs, of community-based surveillance and treatment of cases of severe trachoma (TI) semi-annually or every 4 months?

DETAILED DESCRIPTION:
An important component of a trachoma control program is the effective use of antibiotics, particularly azithromycin, to reduce the pool of chlamydial ocular infection in the communities. A reduction in the pool of infection will reduce the likelihood of transmission and, coupled with effective hygiene and environmental changes, theoretically lead to reduction in disease to the point where active trachoma is no longer a public health problem. Our previous experience with the use of azithromycin for community treatment has shown that even with high rates of coverage, hyperendemic communities will start to experience re-emergent trachoma following treatment by one year. Therefore, it is urgent to determine if there is another treatment strategy for these villages to keep the pool of infection low, and eventually eliminated.A combination approach consisting of mass treatment at yearly intervals and surveillance with a targeted treatment approach in the interim period may be effective in maintaining the low rate of re-emergent disease.We propose to test the cost-effectiveness of three alternative strategies for the frequency of provision of azithromycin, in the context of the Tanzanian National Trachoma Control Program. The strategies have been developed to build on the epidemiological knowledge of trachoma in this area, to be locally appropriate in terms of feasibility and personnel, and to be consistent with the goal of enhancing community control of the program.

A total of nine villages in the Kongwa district of Tanzania will be randomized to one of three groups (a total of three villages per group). The nine villages, with active trachoma rates in pre-school children of 50% or greater, would be slated for enrollment in the National Program, but not currently receiving treatment. Surveys for active trachoma status would be carried out in 300 randomly selected, children ages 1-7 years (pre-school)in each village at baseline, at 6 months post mass treatment, and at one, two, and three years post baseline. The following treatment strategies will be used:

Control villages: Usual practice: The three villages randomized to this arm would receive mass treatment of the community once a year as part of the Tanzania National Trachoma Control program.

Intervention 1. Usual practice plus community surveillance for TI cases and treatment at 6 months: The three villages randomized to this arm would receive mass treatment, similar to the usual practice arm, but in addition, would have a cadre of community volunteers, trained to recognize TI. They will screen their neighborhoods, examining all pre-school children and mothers, and arrange with the health worker for another round of treatment for TI cases and their families at 6 months, and 18 months post baseline.

Intervention 2: Usual practice plus community surveillance for TI cases and treatment every 4 months: The three villages randomized to this arm would have an approach identical to intervention 1, but with surveillance and treatment of TI cases at 4 and 8 months instead of at 6 months.For the second year, they would have surveillance and treatment at 6 months.

Cost data on the community surveillance and treatment program will be collected throughout the first year. Analyses will focus on the additional benefit on reduction in prevalence of trachoma, and ocular C. trachomatis infection, at one, two, and three years of the two alternative strategies, relative to yearly mass treatment alone, and the cost-effectiveness of the three strategies.

ELIGIBILITY:
Inclusion Criteria:

* villages not in the Tanzania National Trachoma control Program in Kongwa, Tanzania
* villages with population size less than 5,000
* sentinel children: ages 1 year to 7 years

Exclusion Criteria:

* Village leadership refuses to allow village participation
* sentinel children: previous history of treatment with azithromycin
* sentinel children: another family member (child)already enrolled in study

Ages: 12 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2700
Dates: Start 2002-04; Study Completion 2005-11

PRIMARY OUTCOMES:
trachoma
ocular C. trachomatis

CONTACTS AND LOCATIONS:
Overall Officials: Sheila K West, Principal Investigator — Johns Hopkins University
Locations (2):
- Johns Hopkins university, Baltimore, Maryland, United States
- Kongwa Trachoma Project, Kongwa, Dodoma, Tanzania